CLINICAL TRIAL: NCT04963075
Title: Non-Invasive Multisensory Rehabilitation of Hemianopia
Brief Title: Multisensory Rehabilitation of Hemianopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Neuroscience Clinical Trial and Innovation Center (NCTIC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00074687
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Hemianopia
Keywords: visual cortex injury; stroke; blindness; cortical damage
MeSH Terms: conditions — Hemianopsia; Stroke; Blindness

STUDY DESIGN:
Intervention Model Description: Subjects will participate in weekly sessions (1.5-2 hours) for three months which contain baseline testing, training, and repeated testing of visual recovery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Unilaterally blind Subjects will be exposed to visual-auditory stimulation (Experimental): The over-arching objective is to evaluate the functional recovery of vision in hemianopic patients engaged with a multisensory training paradigm. Unilaterally blind participants will participate in weekly training sessions in which they are exposed to high-density spatiotemporally congruent and consistent visual-auditory stimulation. The participants will be tested on a battery of visual tasks probing different levels of function in different environments in a longitudinal study to track recovery.
  Interventions: Device: multisensory rehabilitation paradigm

INTERVENTIONS:
Device: multisensory rehabilitation paradigm — In initial ("training") sessions, subjects will be exposed (and respond) to spatiotemporally congruent pairs of visual-auditory stimuli presented within their blinded field, with occasional probes of unisensory visual stimuli on both sides of space. Once recovery of visual responsiveness in the contralesional field is observed, sessions will alternate between "training/testing" and "testing only" sessions in which performance on the visual battery will be re-assessed.

SUMMARY:
The current proposal is to generate "proof of concept" evidence that hemianopia can be successfully rehabilitated in humans when this multisensory rehabilitation paradigm is used.

DETAILED DESCRIPTION:
The over-arching objective is to evaluate the functional recovery of vision in hemianopic patients engaged with a multisensory training paradigm. Unilaterally blind participants will participate in weekly training sessions in which they are exposed to high-density spatiotemporally congruent and consistent visual-auditory stimulation. The participants will be tested on a battery of visual tasks probing different levels of function in different environments in a longitudinal study to track recovery.

ELIGIBILITY:
Inclusion Criteria:

* adults (<85) of either sex
* diagnosis of a stable homonymous hemianopia (>6 months) with absence of hemineglect
* lesion encompassing at least primary visual cortex but sparing parietal cortex
* normal auditory and cognitive function
* willingness to participate in the three month program
* ability to perform the visual discriminations in their intact field

Exclusion Criteria:

* adults (>85)
* normal auditory and cognitive function
* unwilling to participate in the three month program
* inability to perform the visual discriminations in their intact field

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Number of points detected | 3 months
  To assess recovery of function - number of detected visual points in both hemifields (discrete count variable, higher values are "better")
Reaction time | 3 months
  To assess recovery of function - reaction time of visual detection (continuous variable, lower values are "better")
Distance between perceived and actual stimulus location | 3 months
  To assess recovery of function - localization accuracy/error (continuous variable, lower error is "better")
Low-vision visual functioning questionnaire (LV-VFQ-48) | Baseline
  information processing, and visual motor skills) and overall visual ability estimated from difficulty ratings using the 48-item Veterans Affairs Low-Vision Visual Functioning Questionnaire. The difficulty of each item is rated using the ordered response categories (lower is "better"): (1) not difficult, (2) slightly/moderately difficult, (3) extremely difficult, and (4) impossible. Patients were also allowed to respond that they do not perform an activity for nonvisual reasons.
Low-vision visual functioning questionnaire (LV-VFQ-48) | Month 3
  information processing, and visual motor skills) and overall visual ability estimated from difficulty ratings using the 48-item Veterans Affairs Low-Vision Visual Functioning Questionnaire. The difficulty of each item is rated using the ordered response categories (lower is "better"): (1) not difficult, (2) slightly/moderately difficult, (3) extremely difficult, and (4) impossible. Patients were also allowed to respond that they do not perform an activity for nonvisual reasons.
Humphrey visual field test | Baseline
  The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. The Humphrey visual field test can also be used to detect conditions within the optic nerve of the eye, and certain neurological conditions as well. A normal visual field measures about 90 degrees temporally, 50 degrees superiorly and nasally, and 60 degrees inferiorly. (higher scores are better)
Humphrey visual field test | Month 3
  The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. The Humphrey visual field test can also be used to detect conditions within the optic nerve of the eye, and certain neurological conditions as well. A normal visual field measures about 90 degrees temporally, 50 degrees superiorly and nasally, and 60 degrees inferiorly. (higher scores are better)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Rowland, PhD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

DOCUMENTS (1):
  • Informed Consent Form (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04963075/ICF_000.pdf